CLINICAL TRIAL: NCT04527874
Title: Assessment of a Viral Load Result-driven Automated Differentiated Service Delivery Model for Participants Taking Antiretroviral Therapy in Lesotho
Brief Title: Viral Load Triggered ART Care in Lesotho
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P002-20-1.0
Record Dates: First submitted 2020-03-09; First posted 2020-08-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: cluster-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clusters in the intervention arm receive the VITAL intervention (see intervention)
  Interventions: Behavioral: VITAL model
- Control (No Intervention): Clusters in the control arm continue standard of care.

INTERVENTIONS:
Behavioral: VITAL model — The concept of the VITAL, an automated differentiated service delivery model (aDSDM), is to use viral load results, other clinical characteristics (TB screening results and CD4 cell counts, comorbidities) and participants' preference to automatically triage participants into groups requiring different levels of attention and care. Innovatively, triaging of participants will be done automatically making use of a dedicated mobile App and a viral load database platform.
  To ensure effective flow of information and empowerment of patients, viral load results and other relevant information is sent directly to participants' phones, whereas health care providers receive results directly on their study tablet together with the recommended action. Further features of the platform are preference-based tailored adherence reminders and automated calls to participants for symptomatic tuberculosis screening.
  Other Names: automated differentiated service delivery
  Arms: Intervention

SUMMARY:
This cluster randomized clinical trial at 18 nurse-led rural health centers in Lesotho will test an automated differentiated service delivery model using viral load results, other clinical characteristics and participants' preference to automatically triage participants into groups requiring different levels of attention and care.

DETAILED DESCRIPTION:
To sustainably provide good quality care to increasing numbers of people living with HIV (PLHIV) receiving antiretroviral therapy (ART), care delivery has to shift from a "one-size-fits-all" approach to differentiated care models. Such models should reallocate resources from patients who are doing well to patient groups who may need more attention, such as those with treatment failure or medical and psycho-social problems. Ideally, such a reallocation allows health systems and patients to save resources while improving quality of care.

One proposed approach to differentiate care and intensity of monitoring is viral load-driven differentiated service delivery. Reducing the intensity of monitoring in patients with suppressed viral load (VL) and no other clinical problems would substantially reduce the workload at health care facilities and save time and transport cost for patients, thus potentially improve long-term engagement in care. Time and resources saved in patients with suppressed VL and no other clinical problems would allow focusing on those participants with elevated viral load and/or other clinical problems (like tuberculosis, which is the most common cause of mortality among PLHIV in sub-Saharan Africa). This may potentially improve PLHIVs' clinical outcome through intensified adherence support, clinical follow-up and timely switches to second-line ART. In many settings in sub-Saharan Africa, however, the potential of VL monitoring to differentiate care is not exploited and thus constitutes a missed opportunity. In Lesotho it was shown that the majority of unsuppressed VLs are not acted upon in a timely manner, be it due to providers and patients not being aware of the results or health care providers not being proficient in the management of treatment failure.

The concept of the proposed automated differentiated service delivery model (aDSDM) is to use VL results, other clinical characteristics (TB screening results and CD4 cell counts) and participants' preference to automatically triage participants into groups requiring different levels of attention and care. Innovatively, triaging of participants will be done automatically capitalising on an existing VL database platform. The implemented aDSDM will differentiate care according to three elements:

* clinical characteristics (with focus on VL measurement)
* sub-population (women, men)
* participants' and health care providers' preferences

To ensure effective flow of information, VL results and other relevant information is sent directly to participants' phones, whereas health care providers receive results directly on their study tablet together with the recommended action. Further features of the platform are preference-based tailored adherence reminders and automated calls to participants for symptomatic tuberculosis screening. The proposed aDSDM is designed for being scaled up at national and regional level as it mainly builds on automated triage and communication with participants and health care workers, thus not requiring additional human resources.

ELIGIBILITY:
Inclusion criteria:

* nurse-led public or missionary clinic in the districts of Butha-Buthe and Mokhotlong;
* consent of clinic management (signed agreement with clinic management);
* access to the internet (internet connection must not be constant, but there must be possibility to down- and upload information daily); and
* the clinic sends plasma VL samples to Butha-Buthe government hospital laboratory for analysis.

Exclusion criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5809 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Engagement in care with documented viral suppression | 16-28 months after enrollment
  Proportion of participants engaged in care (defined as documented visit attendance) with documented viral suppression (<50 copies/mL) 24 months (16-28 months) after enrollment

SECONDARY OUTCOMES:
Viral re-suppression | 16-28 months after enrollment
  Proportion of participants with viral re-suppression (<50 copies/mL) 24 months (16-28 months) after enrollment among all participants with an unsuppressed VL (≥ 50 copies/mL) during the first 12 months of follow-up
Sustained viral suppression | 16-28 months after enrollment
  Proportion of participants with sustained viral suppression (defined as >1 VL <50 copies/mL) during 24 months (16-28 months) follow-up
Mortality rate | at 12 and 24 months after enrollment
  All-cause mortality
Tuberculosis | at 12 and 24 months after enrollment
  Proportion of participants with confirmed tuberculosis diagnosis
Disengagement from care | at 12 and 24 months after enrollment
  Proportion of participants disengaged from care (defined as no documented visit attendance) at 12 months (8-16 months) and 24 months (16-28 months) after enrollment
Time to follow-up | at 24 months after enrollment
  Time to follow-up viral load in case of an unsuppressed VL (≥50 copies/mL)
Time to ART regimen adaption | at 24 months after enrollment
  Time to ART regimen adaption in case of virologic failure
Rate of clinic visits | at 24 months after enrollment
  Number of clinic visits throughout the study period
Proportion of participants with ART regimen modification | at 12 and 24 months after enrollment
  12. Proportion of participants with ART regimen modification due to virologic failure at 12 and 24 months among participants with virologic failure
Proportion of participants receiving a course of TPT | at 24 months after enrollment
  Proportion of participants having received a course of TPT throughout the study period.

OTHER OUTCOMES:
Proportion of participants requesting a VL result notification through SMS | at 24 months after enrollment
  in intervention clusters
Proportion of SMS delivered successfully | at 24 months after enrollment
  in intervention clusters
Proportion of participants using the call-back option through District ART Nurse | at 24 months after enrollment
  in intervention clusters

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, Prof, Study Chair — University Hospital, Basel, Switzerland
Locations (18):
- Lesotho (18):
  - Boiketsiso Health Center, Butha-Buthe
  - Linakeng Health Center, Butha-Buthe
  - Makhunoane Health Center, Butha-Buthe
  - Motete Health Center, Butha-Buthe
  - Muela Health Center, Butha-Buthe
  - Ngoajane Health Center, Butha-Buthe
  - Rampai Health Center, Butha-Buthe
  - St Paul Health Center, Butha-Buthe
  - St. Peters Health Center, Butha-Buthe
  - Tsime Health Center, Butha-Buthe
  - Libibing, Mokhotlong
  - Linakaneng health center, Mokhotlong
  - Malefiloane health center, Mokhotlong
  - Mapholaneng, Mokhotlong
  - Moeketsane, Mokhotlong
  - Molikaliko health center, Mokhotlong
  - St. James, Mokhotlong
  - St. Martins, Mokhotlong

IPD SHARING:
Plan to Share IPD: Yes
A subset of the key pseudo-anonymised individual participant data collected during the study, along with a data dictionary, will be made available upon request to the Division of Clinical Epidemiology at the University Hospital Basel.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: upon publication of the trial results
Access Criteria: upon request

REFERENCES:
- [Background] Tschumi N, Lerotholi M, Kopo M, Kao M, Lukau B, Nsakala B, Chejane N, Motaboli L, Lee T, Barnabas R, Shapiro AE, van Heerden A, Lejone TI, Amstutz A, Brown JA, Heitner J, Belus JM, Chammartin F, Labhardt ND. Assessment of a viral load result-triggered automated differentiated service delivery model for people taking ART in Lesotho (the VITAL study): Study protocol of a cluster-randomized trial. PLoS One. 2022 May 5;17(5):e0268100. doi: 10.1371/journal.pone.0268100. eCollection 2022. PMID 35511950
- [Derived] Harder MT, Mokete M, Chammartin F, Lerotholi M, Motaboli L, Kopo M, Kao M, Mokebe M, Chejane N, Mahlatsi P, Nyakane M, Tarumbiswa T, Labhardt ND, Tschumi N, Belus JM. Cervical cancer screening delay and associated factors among women with HIV in Lesotho: a mixed-methods study. BMC Womens Health. 2024 Oct 1;24(1):543. doi: 10.1186/s12905-024-03382-8. PMID 39354488

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04527874/SAP_001.pdf